CLINICAL TRIAL: NCT00005045
Title: Phase II Study of Carboxyamidotriazole (CAI, NSC #609974) in Patients With Advanced Renal Cell Carcinoma Refractory to Immunotherapy
Brief Title: Carboxyamidotriazole in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067636; ECOG-4896
Record Dates: First submitted 2000-04-06; First posted 2004-06-09 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2005-12

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — carboxyamido-triazole

INTERVENTIONS:
Drug: carboxyamidotriazole

SUMMARY:
RATIONALE: Carboxyamidotriazole may stop the growth of kidney cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of carboxyamidotriazole in treating patients who have advanced kidney cancer that has not responded to biological therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the disease free progression at 6 months in patients with locally recurrent or metastatic renal cell cancer (refractory to immunotherapy) treated with carboxyamidotriazole. II. Evaluate the progression free survival rate and response rate in these patients on this regimen. III. Evaluate the toxic effect of this regimen on these patients.

OUTLINE: Patients receive oral carboxyamidotriazole daily. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients with stable disease may discontinue therapy after 6 courses. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and every 12 months thereafter until death.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced renal cell cancer Locally recurrent or metastatic lesions not amenable to current resection Progressive disease defined as 25% increase from last measurement or new lesions Bidimensionally measurable disease No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 OR Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGOT and/or SGPT less than 2 times upper limit of normal Renal: Creatinine less than 2.0 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No other serious medical illness or active infection that would preclude chemotherapy compliance No other prior malignancy unless curatively treated and disease free for the past 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy At least 1 (but no more than 2) prior biologic regimen(s) (i.e., interleukin-2, interferon alfa, or combination) and recovered Regimen defined as at least 8 weeks of treatment Prior sargramostim allowed Chemotherapy: No prior chemotherapy Endocrine therapy: At least 4 weeks since prior hormonal therapy (i.e., megestrol or tamoxifen) and recovered Radiotherapy: No prior radiotherapy to study lesions At least 4 weeks since prior radiotherapy and recovered No concurrent palliative radiotherapy Surgery: Prior nephrectomy allowed Recovered from any recent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Friedland, MD, Study Chair — University of Pittsburgh
Locations (55):
- United States (52):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - Kaplan Cancer Center, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny University, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Dutcher JP, Leon L, Manola J, Friedland DM, Roth B, Wilding G; Eastern Cooperative Oncology Group. Phase II study of carboxyamidotriazole in patients with advanced renal cell carcinoma refractory to immunotherapy: E4896, an Eastern Cooperative Oncology Group Study. Cancer. 2005 Dec 1;104(11):2392-9. doi: 10.1002/cncr.21473. PMID 16222691
- [Result] Friedland D, Leon L, Manola J, et al.: Carboxyamidotriazole (CAI) in patients with advanced renal cell cancer (RCC) refractory to immunotherapy: an ECOG phase II trial. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2424, 2002.